CLINICAL TRIAL: NCT02181803
Title: A Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8189 in Healthy Volunteers and in Schizophrenia Patients
Brief Title: MK-8189 Multiple Dose Study in Healthy Volunteers and Schizophrenia Participants (MK-8189-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8189-003
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — MK-8189

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1 Panel A & B MK-8189 Monotherapy 2-40 mg: Schizophrenic (Experimental): Participants with schizophrenia will receive monotherapy of MK-8189 in escalating doses starting at 2 mg once daily (QD) up to 40 mg QD, depending on safety and tolerability
  Interventions: Drug: MK-8189
- Part 2 Panel C MK-8189 Add-on Therapy 2-20 mg: Schizophrenic (Experimental): Participants with schizophrenia will receive add-on therapy of MK-8189 in escalating doses starting at 2 mg QD up to 20 mg QD, depending on safety and tolerability
  Interventions: Drug: MK-8189; Drug: Base Monotherapy
- Part 2 Panel C MK-8189 Add-on Therapy 4-20 mg: Schizophrenic (Experimental): Participants with schizophrenia will receive add-on therapy of MK-8189 in escalating doses starting at 4 mg QD up to 20 mg QD, depending on safety and tolerability
  Interventions: Drug: MK-8189; Drug: Base Monotherapy
- Part 3 Panel D MK-8189 Monotherapy 2-16 mg: Healthy (Experimental): Healthy participants will receive monotherapy of MK-8189 in escalating doses starting at 2 mg QD up to 16 mg QD, depending on safety and tolerability
  Interventions: Drug: MK-8189
- Part 1 Panel A & B Placebo Monotherapy: Schizophrenic (Placebo Comparator): Participants with schizophrenia will receive dose-matched placebo to MK-8189 monotherapy
  Interventions: Drug: Placebo
- Part 2 Panel C Placebo Add-on Therapy: Schizophrenic (Placebo Comparator): Participants with schizophrenia will receive dose-matched placebo to MK-8189 add-on therapy
  Interventions: Drug: Placebo; Drug: Base Monotherapy
- Part 3 Panel D Placebo Monotherapy: Healthy (Placebo Comparator): Healthy participants will receive dose-matched placebo to MK-8189 monotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8189 — MK-8189, oral, 2 mg and/or 10 mg tablets, taken QD for a total daily dose of 2 mg, 4 mg, 8 mg, 10 mg, 12 mg, 14 mg, 16 mg, 20 mg, or 40 mg
  Arms: Part 1 Panel A & B MK-8189 Monotherapy 2-40 mg: Schizophrenic; Part 2 Panel C MK-8189 Add-on Therapy 2-20 mg: Schizophrenic; Part 2 Panel C MK-8189 Add-on Therapy 4-20 mg: Schizophrenic; Part 3 Panel D MK-8189 Monotherapy 2-16 mg: Healthy
Drug: Placebo — Placebo matching oral 2 mg and/or 10 mg MK-8189 tablets, taken QD
  Arms: Part 1 Panel A & B Placebo Monotherapy: Schizophrenic; Part 2 Panel C Placebo Add-on Therapy: Schizophrenic; Part 3 Panel D Placebo Monotherapy: Healthy
Drug: Base Monotherapy — For Part 2 only: participants need to be on monotherapy with an atypical antipsychotic medication (eg, Olanzapine, Quetiapine, Paliperidone, Asenapine, Iloperidone, Aripirprazole, Lurasidone, Risperidone [not to exceed daily dose of 6 mg], or Ziprasidone.) The participant should be on a stable and well tolerated treatment regimen for at least 2 months prior to screening. NOTE: Clozapine is not allowed.
  Arms: Part 2 Panel C MK-8189 Add-on Therapy 2-20 mg: Schizophrenic; Part 2 Panel C MK-8189 Add-on Therapy 4-20 mg: Schizophrenic; Part 2 Panel C Placebo Add-on Therapy: Schizophrenic

SUMMARY:
This 3-part dose titration study will assess MK-8189 safety, tolerability, pharmacokinetics (PK), and central nervous system activity. Part 1 (Panels A and B) will assess MK-8189 administered as monotherapy in participants with schizophrenia. Part 2 (Panel C) will assess MK-8189 administered as add-on to atypical antipsychotic treatment in participants with schizophrenia. Part 3 (Panel D) will assess monotherapy with MK-8189 in healthy participants, including those of Japanese descent. The primary hypothesis is that there is at least one dose of MK-8189 that is generally safe and well-tolerated which will have the desired PK parameters in participants with schizophrenia.

DETAILED DESCRIPTION:
As specified by Phase 1 protocol-flexible language in the protocol, modifications to the dose or dosing regimen can be made to achieve the scientific goals of the trial objectives and/or ensure appropriate safety of the trial participants. The proposed doses for each Part may be adjusted downward based on evaluation of safety, tolerability, and pharmacokinetic data observed in previous panels.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR SCHIZOPHRENIA PARTICIPANTS

* Male or non-pregnant and non-breast feeding female. If participant is male with a female partner of child-bearing potential, participant must agree to use a medically acceptable method of contraception during the trial and for 120 days after the last dose of trial drug. If their partner is pregnant, males must agree to use a condom
* Body Mass Index (BMI) ≥ 18.5 and ≤ 40 kg/m^2
* Meet diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria with the onset of the first episode being no less than 2 years prior to study entry
* Be in the non-acute phase of illness and clinically stable for 3 months prior to screening
* History of receiving and tolerating antipsychotic medication within the usual dose range employed for schizophrenia
* Participants with hypothyroidism, diabetes, high blood pressure, chronic respiratory conditions or other mild forms of these medical conditions could be considered as candidates for study enrollment if their condition is stable and the prescribed dose and regimen of medication is stable for at least 3 months prior to screening and there are no expected changes in comedication during the study
* Has a negative urinary drug screen at screening

INCLUSION CRITERIA FOR HEALTHY PARTICIPANTS

* Male, or non-pregnant and non-breast feeding female of Japanese or non-Japanese descent. If participant is male with a female partner of child-bearing potential, participant must agree to use a medically acceptable method of contraception during the trial and for 120 days after the last dose of trial drug. If their partner is pregnant, males must agree to use a condom
* Body Mass Index (BMI) ≥ 18.5 and ≤ 35 kg/m^2
* In good health
* Nonsmoker and/or has not used nicotine or nicotine-containing products (e.g., nicotine patch) for at least approximately 3 months
* Has a negative urinary drug screen at screening

Exclusion Criteria:

EXCLUSION CRITERIA FOR SCHIZOPHRENIA PARTICIPANTS

* DSM-IV axis I psychiatric diagnosis other than schizophrenia or schizoaffective disorder within one month of screening
* Has evidence or history of mental retardation, borderline personality disorder, anxiety disorder, or organic brain syndrome
* History of neuroleptic malignant syndrome or moderate to severe tardive dyskinesia
* Untreated or uncompensated clinically significant renal, endocrine, hepatic, respiratory, gastrointestinal, psychiatric, neurologic, cardiovascular, hematological, immunological or cerebrovascular disease, malignance, allergic disease or other chronic and/or degenerative process at screening
* Has a history of cancer (malignancy) with certain exceptions
* Treatment with clozapine for schizophrenia or treatment with monoamine oxidase inhibitors within 3 months of screening
* Received a parenteral depot antipsychotic medication within 3 months of screening
* Participated in another investigational study within 4 weeks, prior to screening

EXCLUSION CRITERIA FOR HEALTHY PARTICIPANTS

* History of clinically significant endocrine, gastrointestinal, cardiovascular (including hypertension, angina, coronary artery disease, valvular disease, heart rate or rhythm abnormalities), hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Mentally or legally incapacitated
* History of clinically diagnosed depression, anxiety disorder, or any history of psychiatric disorders having required drug treatment or hospitalization
* History of cancer (malignancy)
* Unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies throughout the trial
* Participated in another investigational study within 4 weeks, prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2015-04-23 (Actual); Study Completion 2015-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-three schizophrenia participants and 12 healthy volunteers were randomized to either MK-8189 or placebo in Part 1 Panels A & B, Part 2 Panel C, or Part 3 Panel D. MK-8189 dose and schedule were modified for participants based on tolerability.
Groups:
- Part 1 Panel A & B MK-8189 Monotherapy 2-4 mg: Schizophrenic: Participant with Schizophrenia received monotherapy of MK-8189 in escalating doses: 2 mg once daily (QD) Days 1-4 and 4 mg QD Days 5-14
- Part 1 Panel A & B MK-8189 Monotherapy 2-12 mg: Schizophrenic: Participants with Schizophrenia received monotherapy of MK-8189 in escalating doses: 2 mg QD Days 1-4, 4 mg QD Days 5-8, 8 mg QD Days 9-11, and 12 mg QD Days 12-14
- Part 1 Panel A & B Placebo Monotherapy: Schizophrenic: Participants with Schizophrenia received dose-matched placebo to MK-8189 monotherapy on Days 1-14
- Part 2 Panel C MK-8189 Add-on Therapy 2-12 mg: Schizophrenic: Participants with Schizophrenia received add-on therapy of MK-8189 in escalating doses: 2 mg QD Days 1-4, 4 mg QD Days 5-8, 8 mg QD Days 9-11, and 12 mg QD Days 12-14
- Part 2 Panel C MK-8189 Add-on Therapy 4-16 mg: Schizophrenic: Participants with Schizophrenia received add-on therapy of MK-8189 in escalating doses: 4 mg QD Days 1-4, 8 mg QD Days 5-8, 12 mg QD Days 9-11, and 16 mg QD Days 12-14
- Part 2 Panel C Placebo Add-on Therapy: Schizophrenic: Participants with Schizophrenia received dose-matched placebo to MK-8189 add-on therapy on Days 1-14
- Part 3 Panel D MK-8189 Monotherapy 2-12 mg: Healthy: Healthy participants received monotherapy of MK-8189 in escalating doses: 2 mg QD Days 1-4, 4 mg QD Days 5-8, 8 mg QD Days 9-11, and 12 mg QD Days 12-14
- Part 3 Panel D MK-8189 Monotherapy 2-8 mg: Healthy: Healthy participant received monotherapy of MK-8189 in escalating doses: 2 mg QD Days 1-4, 4 mg QD Days 5-8, and 8 mg QD days 9-14
- Part 3 Panel D Placebo Monotherapy: Healthy: Healthy participants received dose-matched placebo to MK-8189 monotherapy on Days 1-14
Period: Overall Study
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2-4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 2-12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2-12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4-16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2-12 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 2-8 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Started | 1 | 13 | 4 | 13 | 6 | 6 | 9 | 1 | 2
Completed | 1 | 9 | 4 | 11 | 6 | 6 | 8 | 0 | 2
Not Completed | 0 | 4 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2-4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 2-12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2-12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4-16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2-12 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 2-8 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy | Total
Number analyzed (Participants) | 1 | 13 | 4 | 13 | 6 | 6 | 9 | 1 | 2 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.0 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 44.2 (8.7) | 44.0 (9.0) | 43.8 (8.9) | 41.7 (14.7) | 44.5 (7.6) | 43.3 (8.7) | 55.0 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 43.0 (5.7) | 43.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 6 | 3 | 1 | 2 | 1 | 0 | 17
  Male | 1 | 10 | 3 | 7 | 3 | 5 | 7 | 0 | 2 | 38

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration at 24 Hours Post-dose (C24hr) of MK-8189 in Schizophrenia Participants
Description: C24hr was defined as the concentration of MK-8189 observed in plasma at the 24-hour nominal sampling time after administration of MK-8189. In participants receiving MK-8189, blood samples were collected pre-dose and 24 hours post-dose to estimate C24hr following MK-8189 administration. As specified by the protocol, C24hr was analyzed by part, dose and dosing schedule. Due to differing dosing schedules, some time points were not applicable for certain arms/doses as indicated by zero participants analyzed entered in the table. Per protocol, healthy participants (Part 3) and participants receiving placebo were excluded from C24 analysis.
Time Frame: Day 1, 4, 8, 11 and 14 pre-dose and 24 hours post-dose
Population: Schizophrenia participants who received ≥1 dose of MK-8189, complied with the protocol and had C24 data available for Days 1, 4, 8, 11, or 14. Due to differing dosing schedules, some time points were not applicable for some arms (shown by 0 participants analyzed). Per protocol, healthy participants (Part 3) and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 2 mg QD starting on Day 1 and continuing up to Day 4, based on participant tolerability
- Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 4 mg QD starting on Day 5 and continuing up to Day 14, based on participant tolerability
- Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 8 mg QD starting on day 9 and continuing up to Day 11, based on participant tolerability
- Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic: Participants with Schizophrenia received monotherapy MK-8189 oral dose of 12 mg QD starting on Day 12 and continuing up to Day 14, based on participant tolerability
- Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic: Participants with Schizophrenia received add-on therapy MK-8189 oral dose of 2 mg QD starting on Day 1 and continuing up to Day 4, based on participant tolerability
- Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic: Participants with Schizophrenia received add-on therapy MK-8189 oral dose of 4 mg QD starting on Day 1 and continuing up to Day 8, based on participant tolerability
- Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic: Participants with Schizophrenia received add-on therapy MK-8189 oral dose of 8 mg QD starting on Day 5 and continuing up to Day 11, based on participant tolerability
- Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic: Participants with Schizophrenia received add-on therapy MK-8189 oral dose of 12 mg QD starting on Day 9 and continuing up to Day 14, based on participant tolerability
- Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic: Participants with Schizophrenia received add-on therapy MK-8189 oral dose of 16 mg QD starting on Day 12 and continuing up to day 14, based on participant tolerability
- Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy: Healthy participants received monotherapy MK-8189 oral dose of 2 mg QD starting on Day 1 and continuing up to Day 4, based on participant tolerability
- Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy: Healthy participants received monotherapy MK-8189 oral dose of 4 mg QD starting on Day 5 and continuing up to Day 8, based on participant tolerability
- Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy: Healthy participants received monotherapy MK-8189 oral dose of 8 mg QD starting on Day 9 and continuing up to Day 14, based on participant tolerability
- Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy: Healthy participants received monotherapy MK-8189 oral dose of 12 mg QD starting on Day 12 and continuing up to Day 14, based on participant tolerability
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 13 | 12 | 10 | 9 | 0 | 13 | 11 | 11 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
nM
  Day 1: number analyzed (Participants) | 13 | 0 | 0 | 0 | 0 | 13 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 | 67.0 (31.7) |  |  |  |  | 60.5 (37.1) | 161 (39.8) |  |  |  |  |  |  |  |  |
  Day 4: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4 | 81.1 (94.8) |  |  |  |  | 80.9 (49.1) | 242 (67.9) |  |  |  |  |  |  |  |  |
  Day 8: number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 |  | 183 (52.2) |  |  |  |  | 174 (39.4) | 419 (59.6) |  |  |  |  |  |  |  |
  Day 11: number analyzed (Participants) | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11 |  | 148 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 387 (42.0) |  |  |  |  | 321 (45.1) | 563 (72.3) |  |  |  |  |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 9 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14 |  | 149 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed |  | 459 (33.3) |  |  |  |  | 517 (52.0) | 655 (69.0) |  |  |  |  |  |

2. Primary Outcome: Area Under the Plasma-concentration Curve at Zero to 24 Hours Post-dose (AUC[0-24hr]) of MK-8189 in Schizophrenia Participants
Description: AUC was defined as a measure of MK-8189 exposure that was calculated as the product of plasma drug concentration and time. The linear-up-log down rule was used to estimate AUC. Blood samples were collected pre-dose and up to 24 hours post-dose to estimate AUC(0-24hr) following MK-8189 administration. As specified by the protocol, AUC(0-24hr) was analyzed by part, dose and dosing schedule. Due to differing dosing schedules, some time points were not applicable for certain arms/doses as indicated by zero participants analyzed entered in the table. Per protocol, healthy participants (Part 3) and participants receiving placebo were excluded from AUC(0-24hr) analysis.
Time Frame: Day 1 pre-dose and 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose; Days 4, 8, 11 pre-dose and 6, 10, 16, 24 hours post-dose; Day 14 pre-dose and 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: Schizophrenia participants who received ≥1 dose of MK-8189, complied with the protocol and had AUC(0-24hr) data available for Days 1, 4, 8, 11, or 14. Due to differing dosing schedules, some time points were not applicable for some arms (shown by 0 participants analyzed). Per protocol, healthy participants (Part 3) and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 13 | 12 | 10 | 9 | 0 | 13 | 11 | 11 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
nM*hr
  Day 1: number analyzed (Participants) | 13 | 0 | 0 | 0 | 0 | 13 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 | 1090 (29.8) |  |  |  |  | 1040 (27.3) | 2600 (41.0) |  |  |  |  |  |  |  |  |
  Day 4: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4 | 2160 (69.6) |  |  |  |  | 1810 (42.7) | 5740 (57.8) |  |  |  |  |  |  |  |  |
  Day 8: number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 |  | 4390 (54.4) |  |  |  |  | 4300 (31.5) | 10500 (58.7) |  |  |  |  |  |  |  |
  Day 11: number analyzed (Participants) | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11 |  | 4720 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 9770 (40.8) |  |  |  |  | 8540 (31.2) | 14900 (58.9) |  |  |  |  |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 9 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14 |  | 4100 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed |  | 12300 (27.0) |  |  |  |  | 13200 (38.5) | 18700 (59.4) |  |  |  |  |  |

3. Primary Outcome: Maximum Observed Post-dose Plasma Concentration (Cmax) of MK-8189 in Schizophrenia Participants
Description: Cmax was defined as the maximum concentration of MK-8189 observed in plasma. Blood samples were collected pre-dose and up to 48 hours post-dose at multiple time points to estimate Cmax following MK-8189 administration. As specified by the protocol, Cmax was analyzed by part, dose and dosing schedule. Due to differing dosing schedules, some time points were not applicable for certain arms/doses as indicated by zero participants analyzed entered in the table. Per protocol, healthy participants (Part 3) and participants receiving placebo were excluded from Cmax analysis.
Time Frame: Day 1 pre-dose and 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post-dose; Days 4, 8, 11 pre-dose and 6, 10, 16, 24 hours post-dose; Day 14 pre-dose and 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 36, 48 hours post-dose
Population: Schizophrenia participants who received ≥1 dose of MK-8189, complied with the protocol and had Cmax data available for Days 1, 4, 8, 11, or 14. Due to differing dosing schedules, some time points were not applicable for some arms (shown by 0 participants analyzed). Per protocol, healthy participants (Part 3) and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 13 | 12 | 10 | 9 | 0 | 13 | 11 | 11 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
nM
  Day 1: number analyzed (Participants) | 13 | 0 | 0 | 0 | 0 | 13 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 | 70.7 (29.9) |  |  |  |  | 63.6 (27.5) | 165 (39.9) |  |  |  |  |  |  |  |  |
  Day 4: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4 | 118 (60.7) |  |  |  |  | 90.6 (41.7) | 277 (59.7) |  |  |  |  |  |  |  |  |
  Day 8: number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 |  | 212 (52.0) |  |  |  |  | 210 (29.8) | 518 (56.5) |  |  |  |  |  |  |  |
  Day 11: number analyzed (Participants) | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11 |  | 285 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed | 472 (40.8) |  |  |  |  | 409 (28.8) | 718 (53.4) |  |  |  |  |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 9 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14 |  | 209 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed |  | 628 (28.5) |  |  |  |  | 638 (34.8) | 1050 (46.3) |  |  |  |  |  |

4. Primary Outcome: Time Post-dose at Which the Maximum Plasma Concentration (Tmax) of MK-8189 Was Observed in Schizophrenia Participants
Description: Tmax was defined as the time required post dose to reach a maximum plasma concentration of MK-8189. It was estimated as the actual sampling time at the highest MK-8189 plasma concentration. Blood samples were collected pre-dose and up to 48 hours post-dose at multiple time points to estimate Tmax following MK-8189 administration. As specified by the protocol, Tmax was analyzed by part, dose and dosing schedule. Due to differing dosing schedules, some time points were not applicable for certain arms/doses as indicated by zero participants analyzed entered in the table. Per protocol, healthy participants (Part 3) and participants receiving placebo were excluded from Tmax analysis.
Time Frame: as for outcome 3
Population: Schizophrenia participants who received ≥1 dose of MK-8189, complied with the protocol and had Tmax data available for Days 1, 4, 8, 11, or 14. Due to differing dosing schedules, some time points were not applicable for some arms (shown by 0 participants analyzed). Per protocol, healthy participants (Part 3) and placebo arms were excluded.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 13 | 12 | 10 | 9 | 0 | 13 | 11 | 11 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr
  Day 1: number analyzed (Participants) | 13 | 0 | 0 | 0 | 0 | 13 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 | 20 [12 to 23.83] |  |  |  |  | 23.83 [10.10 to 25.27] | 23.83 [16 to 23.83] |  |  |  |  |  |  |  |  |
  Day 4: number analyzed (Participants) | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 4 | 10 [0 to 23.87] |  |  |  |  | 23.83 [6 to 23.92] | 8 [0 to 23.83] |  |  |  |  |  |  |  |  |
  Day 8: number analyzed (Participants) | 0 | 12 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 |  | 10 [0 to 23.98] |  |  |  |  | 16 [0 to 23.83] | 0 [0 to 10] |  |  |  |  |  |  |  |
  Day 11: number analyzed (Participants) | 0 | 1 | 10 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11 |  | 10 [NA to NA] — Measure of dispersion could not be estimated due to low number of participants analyzed | 10.03 [10 to 23.83] |  |  |  |  | 16 [0 to 23.83] | 16 [6 to 23.83] |  |  |  |  |  |  |
  Day 14: number analyzed (Participants) | 0 | 1 | 0 | 9 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14 |  | 20 [NA to NA] — Measure of dispersion could not be estimated due to low number of participants analyzed |  | 16 [6 to 24] |  |  |  |  | 12 [4 to 20] | 8 [2 to 12] |  |  |  |  |  |

5. Primary Outcome: Time Required for Plasma Concentration of MK-8189 to Decrease by Half (Apparent t1/2) in Schizophrenia Participants on Day 14
Description: t1/2 was defined as the time required to divide the MK-8189 plasma concentration by half after reaching pseudo-equilibrium. At least three quantifiable post-Cmax, terminal phase concentrations collected were used to calculate the apparent t1/2. Blood samples were collected pre-dose and up to 48 hours post-dose at multiple time points on Day 14 to estimate t1/2 following MK-8189 administration. As specified by the protocol, t1/2 was analyzed by part, dose and dosing schedule. Due to differing dosing schedules, the Day 14 timepoint was not applicable for certain arms/doses as indicated by zero participants analyzed entered in the table. Per protocol, healthy participants (Part 3) and participants receiving placebo were excluded from t1/2 analysis.
Time Frame: Day 14 pre-dose and 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 36, 48 hours post-dose
Population: Schizophrenia participants who received ≥1 dose of MK-8189, complied with the protocol and had t1/2 data available for Day 14. Due to differing dosing schedules, some time points were not applicable for some arms/doses (indicated by zero participants analyzed). Per protocol healthy participants (Part 3) and placebo arms were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 0 | 1 | 0 | 8 | 0 | 0 | 0 | 0 | 11 | 6 | 0 | 0 | 0 | 0 | 0 | 0
hr |  | 9.14 (NA) — Measure of dispersion could not be estimated due to low number of participants analyzed |  | 8.38 (37.8) |  |  |  |  | 8.86 (37.4) | 10.4 (43.6) |  |  |  |  |  |

6. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced at least one AE were reported.
Time Frame: Up to Day 28
Population: All participants who received as least one dose of the investigational drug. Per protocol, safety was assessed by part and dose.
Measure: Number; unit: Participants
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 14 | 12 | 10 | 10 | 4 | 13 | 17 | 17 | 17 | 6 | 6 | 10 | 10 | 10 | 9 | 2
Participants | 8 | 6 | 2 | 6 | 3 | 3 | 6 | 7 | 7 | 2 | 4 | 5 | 5 | 6 | 3 | 2

7. Primary Outcome: Number of Participants Who Discontinue From Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to Day 14
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 14 | 12 | 10 | 10 | 4 | 13 | 17 | 17 | 17 | 6 | 6 | 10 | 10 | 10 | 9 | 2
Participants | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

8. Secondary Outcome: Change From Baseline at Day 13 in Mismatched Negativity (MMN) Peak Amplitude in Monotherapy MK-8189-treated Schizophrenia Participants
Description: MMN is a response to deviant tone (stimuli) measured in electroencephalogram (EEG) signals. Difference in deviant EEG waveform amplitude from standard amplitude over time indicates MMN; this difference at peak waveform is MMN peak amplitude. Schizophrenic participants show reduced response to deviant stimuli. Peak amplitude change from baseline (Day -1) to Day 13 was reported. A higher change indicates improved response to deviant stimuli. Scalp EEG signals were collected using a standard system array of 19 electrodes denoted by nomenclature of scalp placement: C3, C4, Cz, F3, F4, F7, F8, Fp1, Fp2, Fz, O1, O2, P3, P4, Pz, T3, T4, T5, T6. As specified by the protocol, MK-8189 add-on therapy schizophrenia participants (Part 2), healthy participants (Part 3) and all placebo-treated participants were excluded from MMN analyses. Per protocol, MMN analyses were planned and executed in all schizophrenia participants receiving MK-8189 monotherapy, irrespective of different dosing schedules.
Time Frame: Baseline and Day 13
Population: Per protocol, MMN analyses were planned and executed in all Schizophrenia participants receiving MK-8189 monotherapy (irrespective of dosing schedule) with EEG electrode data available. Per protocol MK-8189 add-on therapy schizophrenia participants (Part 2), healthy participants (Part 3) and all placebo-treated participants were excluded.
Measure: Mean (95% Confidence Interval); unit: µV
Groups:
- Part 1 Panel A & B MK-8189 Monotherapy 2-12 mg: Schizophrenic: Participants received MK-8189 escalating doses: 2 mg QD Days 1-4, 4 mg QD Days 5-8, 8 mg QD Days 9-11, and 12 mg QD Days 12-14 or alternatively 2 mg QD Days 1-4 and 4 mg QD Days 5-14
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2-12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2-12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4-16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2-12 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 2-8 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
µV
  C3 | 0.959 [-0.218 to 2.137] |  |  |  |  |  |  |
  C4 | 0.812 [-0.169 to 1.794] |  |  |  |  |  |  |
  Cz | 1.170 [-0.203 to 2.543] |  |  |  |  |  |  |
  F3 | 1.547 [0.171 to 2.922] |  |  |  |  |  |  |
  F4 | 1.240 [-0.006 to 2.487] |  |  |  |  |  |  |
  F7 | 0.616 [-0.471 to 1.702] |  |  |  |  |  |  |
  F8 | 0.488 [-1.113 to 2.088] |  |  |  |  |  |  |
  Fp1 | 0.779 [-0.586 to 2.144] |  |  |  |  |  |  |
  Fp2 | 1.103 [-0.480 to 2.687] |  |  |  |  |  |  |
  Fz | 1.462 [0.256 to 2.667] |  |  |  |  |  |  |
  O1 | -0.099 [-1.548 to 1.350] |  |  |  |  |  |  |
  O2 | -0.014 [-1.186 to 1.159] |  |  |  |  |  |  |
  P3 | 0.236 [-1.188 to 1.660] |  |  |  |  |  |  |
  P4 | -0.037 [-1.233 to 1.159] |  |  |  |  |  |  |
  Pz | 0.599 [-0.675 to 1.873] |  |  |  |  |  |  |
  T3 | 1.018 [-1.924 to 3.960] |  |  |  |  |  |  |
  T4 | 0.306 [-2.667 to 3.278] |  |  |  |  |  |  |
  T5 | -0.260 [-3.475 to 2.955] |  |  |  |  |  |  |
  T6 | 0.178 [-2.378 to 2.734] |  |  |  |  |  |  |

9. Secondary Outcome: Change From Baseline at Day 13 in Mismatched Negativity (MMN) Area Under Curve (AUC) in Monotherapy MK-8189-treated Schizophrenia Participants
Description: MMN is a response to deviant tone (stimuli) measured in EEG signals. Difference in deviant EEG waveform amplitude from standard amplitude over time indicates MMN; AUC was measured as the product of MMN amplitude and time. Schizophrenic participants show reduced response to deviant stimuli. AUC change from baseline (Day -1) to Day 13 was reported. A higher change indicates improved response to deviant stimuli. Scalp EEG signals were collected using a standard system array of 19 electrodes denoted by nomenclature of scalp placement: C3, C4, Cz, F3, F4, F7, F8, Fp1, Fp2, Fz, O1, O2, P3, P4, Pz, T3, T4, T5, T6. As specified by the protocol, MK-8189 add-on therapy schizophrenia participants (Part 2), healthy participants (Part 3), and all placebo-treated participants were excluded from MMN analyses. Per protocol, MMN analyses were planned and executed in all schizophrenia participants receiving MK-8189 monotherapy, irrespective of different dosing schedules.
Time Frame: Baseline and Day 13
Population: Per protocol, MMN analyses were planned and executed in all Schizophrenia participants receiving MK-8189 monotherapy (irrespective of dosing schedule) with EEG electrode data available. Per protocol, MK-8189 add-on therapy schizophrenia participants (Part 2), healthy participants (Part 3), and all placebo-treated participants were excluded.
Measure: Mean (95% Confidence Interval); unit: µV*msec
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2-12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2-12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4-16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2-12 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 2-8 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy
Number analyzed (Participants) | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
µV*msec
  C3 | -4.162 [-25.187 to 16.863] |  |  |  |  |  |  |
  C4 | 2.800 [-12.255 to 17.856] |  |  |  |  |  |  |
  Cz | 2.813 [-19.664 to 25.290] |  |  |  |  |  |  |
  F3 | 6.277 [-12.012 to 24.565] |  |  |  |  |  |  |
  F4 | 9.814 [-5.671 to 25.299] |  |  |  |  |  |  |
  F7 | -0.582 [-8.968 to 7.803] |  |  |  |  |  |  |
  F8 | 8.817 [-3.836 to 21.470] |  |  |  |  |  |  |
  Fp1 | 8.390 [-7.696 to 24.476] |  |  |  |  |  |  |
  Fp2 | 11.483 [-9.046 to 32.012] |  |  |  |  |  |  |
  Fz | 7.880 [-14.368 to 30.129] |  |  |  |  |  |  |
  O1 | -3.011 [-23.898 to 17.875] |  |  |  |  |  |  |
  O2 | -10.261 [-24.940 to 4.419] |  |  |  |  |  |  |
  P3 | -9.560 [-34.188 to 15.069] |  |  |  |  |  |  |
  P4 | -9.154 [-29.863 to 11.555] |  |  |  |  |  |  |
  Pz | -10.019 [-36.607 to 16.570] |  |  |  |  |  |  |
  T3 | -15.594 [-48.553 to 17.365] |  |  |  |  |  |  |
  T4 | -3.341 [-23.264 to 16.582] |  |  |  |  |  |  |
  T5 | -19.394 [-47.983 to 9.194] |  |  |  |  |  |  |
  T6 | -12.686 [-39.170 to 13.799] |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Up to Day 28; all-cause mortality was assessed for up to ~9 months
Description: Safety was assessed by part and dose, in all participants who received as least one dose of the investigational drug. Post Study AEs were pooled across the arms in each part of the study. AEs that occurred beyond 14 days of dosing were considered Post Study AEs.
Groups:
- Part 1 Panel A & B Post Study: Schizophrenic: Participants with Schizophrenia who received monotherapy MK-8189 or matching placebo during the treatment period, were followed for safety during the post study period
- Part 2 Panel C Post Study: Schizophrenic: Participants with Schizophrenia who received add-on therapy MK-8189 or matching placebo during the treatment period, were followed for safety during the post study period
- Part 1 Panel D Post Study: Healthy: Healthy participants who received monotherapy MK-8189 or matching placebo during the treatment period, were followed for safety during the post study period
Arm/Group | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic | Part 1 Panel A & B Post Study: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic | Part 2 Panel C Post Study: Schizophrenic | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy | Part 3 Panel D Placebo Monotherapy: Healthy | Part 1 Panel D Post Study: Healthy
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12 | 0/10 | 0/10 | 0/4 | 0/18 | 0/13 | 0/17 | 0/17 | 0/17 | 0/6 | 0/6 | 0/25 | 0/10 | 0/10 | 0/10 | 0/9 | 0/2 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/10 | 0/10 | 0/4 | 0/18 | 0/13 | 0/17 | 0/17 | 0/17 | 0/6 | 0/6 | 0/25 | 0/10 | 0/10 | 0/10 | 1/9 | 0/2 | 0/12
Other Adverse Events (participants affected / at risk) | 8/14 | 6/12 | 2/10 | 6/10 | 3/4 | 0/18 | 3/13 | 6/17 | 7/17 | 7/17 | 2/6 | 4/6 | 1/25 | 5/10 | 5/10 | 6/10 | 2/9 | 2/2 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic (N=14) | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic (N=12) | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic (N=10) | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic (N=10) | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic (N=4) | Part 1 Panel A & B Post Study: Schizophrenic (N=18) | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic (N=13) | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic (N=17) | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic (N=17) | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic (N=17) | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic (N=6) | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic (N=6) | Part 2 Panel C Post Study: Schizophrenic (N=25) | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy (N=10) | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy (N=10) | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy (N=10) | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy (N=9) | Part 3 Panel D Placebo Monotherapy: Healthy (N=2) | Part 1 Panel D Post Study: Healthy (N=12)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Panel A & B MK-8189 Monotherapy 2 mg: Schizophrenic (N=14) | Part 1 Panel A & B MK-8189 Monotherapy 4 mg: Schizophrenic (N=12) | Part 1 Panel A & B MK-8189 Monotherapy 8 mg: Schizophrenic (N=10) | Part 1 Panel A & B MK-8189 Monotherapy 12 mg: Schizophrenic (N=10) | Part 1 Panel A & B Placebo Monotherapy: Schizophrenic (N=4) | Part 1 Panel A & B Post Study: Schizophrenic (N=18) | Part 2 Panel C MK-8189 Add-on Therapy 2 mg: Schizophrenic (N=13) | Part 2 Panel C MK-8189 Add-on Therapy 4 mg: Schizophrenic (N=17) | Part 2 Panel C MK-8189 Add-on Therapy 8 mg: Schizophrenic (N=17) | Part 2 Panel C MK-8189 Add-on Therapy 12 mg: Schizophrenic (N=17) | Part 2 Panel C MK-8189 Add-on Therapy 16 mg: Schizophrenic (N=6) | Part 2 Panel C Placebo Add-on Therapy: Schizophrenic (N=6) | Part 2 Panel C Post Study: Schizophrenic (N=25) | Part 3 Panel D MK-8189 Monotherapy 2 mg: Healthy (N=10) | Part 3 Panel D MK-8189 Monotherapy 4 mg: Healthy (N=10) | Part 3 Panel D MK-8189 Monotherapy 8 mg: Healthy (N=10) | Part 3 Panel D MK-8189 Monotherapy 12 mg: Healthy (N=9) | Part 3 Panel D Placebo Monotherapy: Healthy (N=2) | Part 1 Panel D Post Study: Healthy (N=12)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oromandibular dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Spasmodic dysphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anhedonia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depersonalisation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Derealisation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There were some missing event markers in EEG recordings during data collection, these were imputed for the MMN analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.